CLINICAL TRIAL: NCT02365298
Title: Clinical and Laboratory Study of Lysozyme Deposition on Daily Disposable Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: CR-5695
Record Dates: First submitted 2015-01-22; First posted 2015-02-18 (Estimated); Results first posted 2017-07-13 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-04

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- etafilcon A (Experimental): Worn in a daily disposable modality
  Interventions: Device: etafilcon A; Device: nelfilcon A
- nelfilcon A (Active Comparator): Worn in a daily disposable modality
  Interventions: Device: etafilcon A; Device: nelfilcon A

INTERVENTIONS:
Device: etafilcon A — etafilcon A soft contact lens
  Other Names: Marketed Investigational Soft Contact Lens
Device: nelfilcon A — nelfilcon A
  Other Names: Marketed Investigational Soft Contact Lens

SUMMARY:
In vitro studies show that some hydrogel materials uptake more lysozyme than other hydrogel materials and that this protein remains largely active and promotes reduced cytokine response in an in vitro culture of human corneal epithelial cells. This study investigates whether these data transfer to the in vivo situation.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must read, understand, and sign the Statement of Informed Consent and receive a fully executed copy of the form.
2. The subject must appear able and willing to adhere to the instructions set forth in the clinical protocol.
3. The subject must be willing to follow instructions and maintain the appointment schedule.
4. The subject must be between 18 and 40 years of age (inclusive).
5. The subject's vertex corrected spherical equivalent distance refraction must be in the range of -0.50D to -6.00D in each eye (inclusive).
6. The subject's refractive cylinder must not exceed -1.25DC in each eye after vertexing to the corneal plane.
7. The subject must be a current wearer of spherical, soft contact lenses (no toric, bifocal or multifocal contact lenses, no extended wear or monovision) for at least 5 days/week and at least 8 hours/day during to month prior to enrollment.
8. The subject must own a wearable pair of spectacles and wear them the day of the initial visit.
9. The subject must be an existing wearer of spherical soft contact lenses in both eyes.
10. The subject must have normal eye (i.e., no ocular medications or infections of any type).
11. The subject must be able to wear the study lenses for a minimum seven hours per day.

Exclusion Criteria:

1. Any ocular or systemic allergies or diseases that may interfere with contact lens wear (at the investigator's discretion).
2. Any systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear (at the investigator's discretion).
3. Currently pregnant or lactating (subjects who become pregnant during the study will be discontinued).
4. Any infectious disease (e.g., hepatitis, tuberculosis) or a contagious immunosuppressive disease.
5. Any active ocular infection.
6. Is using any topical medication including artificial tears (ATS) up to two weeks prior to the screening visit.
7. Any participants whose habitual contact lenses are used as an extended wear regimen.
8. Entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or moderate or above corneal distortion by keratometry.
9. Clinically significant (grade 3 or 4) corneal edema, corneal vascularization, corneal staining, or any other abnormalities of the cornea which would contraindicate contact lens wear; clinically significant (grade 3 or 4) tarsal abnormalities or bulbar injection which might interfere with contact lens wear.
10. Any know hypersensitivity or allergic reaction to study products.
11. Participation in any contact lens or lens care product clinical trial within seven days prior to study enrollment.
12. Employee or family member of the Center for Contact Lens Research (e.g., Investigator, Coordinator, Technician).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2015-06-01 (Actual); Study Completion 2015-06-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Waterloo, Waterloo, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Etafilcon a /Nelfilcon A: Subjects that were randomized to receive the etafilcon A lens first, and then to receive the nelfilcon A lens second.
- Nelfilcon A / Etafilcon A: Subjects that were randomized to receive the nelfilcon A lens first, and then to receive the etafilcon A lens second.
Period: Period 1
Arm/Group | Etafilcon a /Nelfilcon A | Nelfilcon A / Etafilcon A
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Etafilcon a /Nelfilcon A | Nelfilcon A / Etafilcon A
Started | 14 | 14
Completed | 12 | 12
Not Completed | 2 | 2
Not completed — incorrect Rx dispensed | 1 | 0
Not completed — Discontinued at request of Sponsor | 1 | 0
Not completed — Test Article longer available | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: All subjects dispensed at least one study lens during the duration of the study.
Groups:
- All Dispensed Subjects: All subjects that were dispensed a study lens.
Arm/Group | All Dispensed Subjects
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.3 (4.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 10
  White | 18
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 28

OUTCOME MEASURES:

1. Primary Outcome: Total Protein and Total Lysosome Deposits
Description: Measurement will be taken after the subject has worn the lenses for a full seven hours
Time Frame: 2 wks after baseline
Population: All subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: (ug/lens)
Groups:
- Etafilcon A: Subjects that wore the etafilcon A lens in either the first or second period of the study.
- Nelfilcon A: Subjects that wore the nelfilcon A lens in either the first or second period of the study.
Arm/Group | Etafilcon A | Nelfilcon A
Number analyzed (Participants) | 24 | 24
(ug/lens)
  Total Lysozyme | 294.58 (113.855) | 1.68 (0.975)
  Active Lysozyme | 244.00 (87.325) | 0.93 (0.650)
  Total Proteins | 482.06 (139.196) | 6.46 (3.953)

2. Primary Outcome: Total Protein and Total Lysosome Deposits
Description: Measurement will be taken after the subject has worn the lenses for a full seven hours
Time Frame: 6 wks after baseline
Population: Subjects that completed all study visits without a major protocol deviation. During the 2nd period subjects continued wearing the current lens that they were randomized to for an additional 6 weeks of wear.
Measure: Mean (Standard Deviation); unit: (ug/lens)
Arm/Group | Etafilcon A | Nelfilcon A
Number analyzed (Participants) | 12 | 11
(ug/lens)
  Total Lysozyme | 349.00 (58.845) | 2.26 (1.460)
  Active Lysozyme | 263.92 (38.562) | 1.13 (0.538)
  Total Proteins | 473.58 (131.432) | 7.46 (4.151)

3. Primary Outcome: Total Protein and Lysosome Deposits
Description: Measurement will be taken after the subject has worn the lenses for a full seven hours
Time Frame: 12 wks after baseline
Population: All subjects that completed all study visits without a major protocol deviation.During the 2nd period subjects continued wearing the current lens that they were randomized to for an additional 6 weeks of wear.
Measure: Mean (Standard Deviation); unit: (ug/lens)
Arm/Group | Etafilcon A | Nelfilcon A
Number analyzed (Participants) | 12 | 12
(ug/lens)
  Total Lysozyme | 289.17 (78.838) | 1.58 (0.851)
  Active Lysozymes | 242.75 (57.974) | 1.01 (0.567)
  Total Proteins | 394.42 (122.302) | 5.87 (3.181)

4. Primary Outcome: Quantity of Cytokines and Albumin in Tear Fluid
Description: Measured cytokines: IL-1β, IL-2, IL-6, IL-8, IL-10, IL-12, IL-13, and TNF-alpha Measurement will be taken after the subject has worn the lenses for a full seven hours.
Time Frame: 2 wks after baseline
Population: Subjects that completed all study visits without a major protocol deviation. All 24 subjects completed the study, however in some subjects the concentration of cytokine levels were below detectable limits in the tear film sample and could not be analyzed.
Measure: Mean (Standard Deviation); unit: (pg/ml)
Arm/Group | Etafilcon A | Nelfilcon A
Number analyzed (Participants) | 23 | 24
(pg/ml)
  TFN-a: number analyzed (Participants) | 10 | 10
  TFN-a | 1.20 (0.528) | 1.17 (1.095)
  IL-1B: number analyzed (Participants) | 13 | 14
  IL-1B | 1.70 (1.810) | 2.32 (3.023)
  IL-2: number analyzed (Participants) | 12 | 10
  IL-2 | 1.19 (0.841) | 1.49 (1.770)
  IL-6: number analyzed (Participants) | 21 | 21
  IL-6 | 12.32 (11.756) | 15.03 (18.835)
  IL-8 | 466.32 (291.109) | 472.91 (273.444)
  IL-10: number analyzed (Participants) | 20 | 19
  IL-10 | 2.02 (1.879) | 1.64 (1.389)
  IL-12: number analyzed (Participants) | 13 | 9
  IL-12 | 2.72 (5.218) | 2.25 (2.685)
  IL-13: number analyzed (Participants) | 12 | 15
  IL-13 | 29.62 (19.510) | 27.23 (23.651)

5. Primary Outcome: Quantity of Cytokines and Albumin in Tear Fluid
Description: Measured cytokines: IL-1β, IL-2, IL-6, IL-8, IL-10, IL-12, IL-13, and TNF-alpha. Measurement will be taken after the subject has worn the lenses for a full seven hours. During the 2nd period subjects continued wearing the current lens that they were randomized to for an additional 6 weeks of wear.
Time Frame: 6 wks after baseline
Population: All subjects that completed all study visits without a major protocol deviation. All 12 subjects completed the study, however in some subjects the concentration of cytokine levels were below detectable limits in the tear film sample and could not be analyzed.
Measure: Mean (Standard Deviation); unit: (pg/ml)
Arm/Group | Etafilcon A | Nelfilcon A
Number analyzed (Participants) | 12 | 12
(pg/ml)
  TNF-a: number analyzed (Participants) | 3 | 4
  TNF-a | 1.20 (1.111) | 0.49 (0.242)
  IL-1B: number analyzed (Participants) | 3 | 3
  IL-1B | 2.83 (1.595) | 4.99 (6.297)
  IL-2: number analyzed (Participants) | 12 | 9
  IL-2 | 1.50 (1.528) | 1.06 (0.569)
  IL-6: number analyzed (Participants) | 11 | 11
  IL-6 | 12.70 (11.281) | 11.91 (17.135)
  IL-8: number analyzed (Participants) | 12 | 11
  IL-8 | 480.99 (353.994) | 481.08 (346.982)
  IL-10: number analyzed (Participants) | 10 | 9
  IL-10 | 0.90 (1.002) | 0.55 (0.341)
  IL-12: number analyzed (Participants) | 4 | 6
  IL-12 | 0.42 (0.139) | 0.56 (0.222)
  IL-13: number analyzed (Participants) | 2 | 2
  IL-13 | 17.78 (17.396) | 14.10 (8.998)

6. Primary Outcome: Quantity of Cytokines and Albumin in Tear Fluid
Description: as for outcome 5
Time Frame: 12 wks after baseline
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: (pg/ml)
Arm/Group | Etafilcon A | Nelfilcon A
Number analyzed (Participants) | 12 | 12
(pg/ml)
  TFN-a: number analyzed (Participants) | 6 | 6
  TFN-a | 0.57 (0.411) | 0.85 (0.772)
  IL-1B: number analyzed (Participants) | 7 | 8
  IL-1B | 5.18 (6.079) | 8.14 (10.250)
  IL-2: number analyzed (Participants) | 8 | 8
  IL-2 | 1.43 (1.314) | 1.09 (0.479)
  IL-6 | 10.18 (6.155) | 21.33 (26.329)
  IL-8: number analyzed (Participants) | 11 | 12
  IL-8 | 473.86 (164.445) | 879.82 (922.383)
  IL-10: number analyzed (Participants) | 6 | 5
  IL-10 | 0.85 (1.060) | 1.17 (0.618)
  IL-12: number analyzed (Participants) | 4 | 3
  IL-12 | 0.74 (0.211) | 0.51 (0.429)
  IL-13: number analyzed (Participants) | 5 | 4
  IL-13 | 14.56 (5.053) | 29.91 (8.963)

ADVERSE EVENTS:
Time Frame: Approximately 81-87 days per subject.
Arm/Group | Etafilcon A | Nelfilcon A
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 0/28 | 2/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etafilcon A (N=28) | Nelfilcon A (N=28)
Common Cold (Infections and infestations) | 0 (0) | 2 (2) — Not Study Related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days